CLINICAL TRIAL: NCT00160342
Title: A Multi-Center, Double-Blind, Placebo-Controlled Comparison of Multiple Doses of Esterified Estrogens and Methyltestosterone, in Combination and Alone, in Relieving Vasomotor Symptoms in Postmenopausal Women
Brief Title: Comparison of Estrogen and Methyltestosterone Combination Treatments for Postmenopausal Hot Flushes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Sheri Rhodes, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S030.2.112; 2005-002887-27
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Hot Flushes, Menopause, Postmenopause
Keywords: Hormone replacement therapy, hot flushes, postmenopause
MeSH Terms: conditions — Hot Flashes | interventions — Estrogens, Esterified (USP); Methyltestosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1 (Active Comparator)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 2 (Experimental)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 3 (Experimental)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 4 (Active Comparator)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 5 (Experimental)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 6 (Experimental)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 7 (Active Comparator)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 8 (Active Comparator)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)
- 9 (Placebo Comparator)
  Interventions: Drug: Esterified Estrogens (EE) and Methyltestosterone (MT)

INTERVENTIONS:
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.15 EE/0.15 MT
  Arms: 1
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.15 EE/0.15 MT
  Arms: 2
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.15 EE/0.30 MT
  Arms: 3
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.30 EE/0.30 MT
  Arms: 5
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.30 EE
  Arms: 4
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.30 EE/0.60 MT
  Arms: 6
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.45 EE
  Arms: 7
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, 0.60 MT
  Arms: 8
Drug: Esterified Estrogens (EE) and Methyltestosterone (MT) — oral tablet, QD, 12 weeks, Placebo
  Arms: 9

SUMMARY:
This is a research study to evaluate the effectiveness, safety and side effects of several dose levels of esterified estrogens (EE) and methyltestosterone (MT) given individually and in combination compared to a placebo (a tablet with no active drug in it) as a possible treatment for vasomotor symptoms (such as hot flushes and flushing) of menopause. EE and testosterone are two hormones which are typically deficient in menopausal women

ELIGIBILITY:
Inclusion Criteria:

1. Be able to communicate with the Investigator and study staff and be able to complete the required study procedures,
2. Be a female of any race between the ages of 45-65 years, in generally good health,
3. Be either naturally or surgically postmenopausal (with or without a uterus)

Exclusion Criteria:

1. Known sensitivity or contraindications to natural or synthetic estrogens, androgens or progestins,
2. History of or current diagnosis of malignant melanoma, breast cancer or any cancer (except non-melanomatous skin cancer) diagnosed less than 5 years prior to beginning the study

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1251 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mean change in frequency of moderate to severe vasomotor symptoms (VMS) from baseline to Week 4 | 4 weeks
Mean change in frequency of moderate to severe VMS from baseline to Week 12 | 12 weeks
Mean change in severity of moderate to severe VMS from baseline to Week 4 | 4 weeks
Mean change in severity of moderate to severe VMS from baseline to Week 12 | 12 weeks

SECONDARY OUTCOMES:
Frequency and severity of moderate to severe and all hot flushes at each week | 12 weeks
Mean change from baseline to Week 12 in the moderate to severe vulvar and vaginal atrophy symptom identified by the subject as most bothersome | 12 weeks
Mean change from baseline to Week 12 in vaginal pH | 12 weeks
Mean change from baseline to Week 12 in vaginal maturation index (parabasal and superficial cells) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (125):
- United States (88):
  - Site 37, Montgomery, Alabama
  - Site 69, Montgomery, Alabama
  - Site 44, Tucson, Arizona
  - Site 6, Jonesboro, Arkansas
  - Site 62, Little Rock, Arkansas
  - Site 70, Carmichael, California
  - Site 85, Carmichael, California
  - Site 87, Northridge, California
  - Site 18, San Diego, California
  - Site 27, San Diego, California
  - Site 54, San Diego, California
  - Site 31, Vista, California
  - Site 68, Walnut Creek, California
  - Site 66, Denver, Colorado
  - Site 4, Groton, Connecticut
  - Site 35, New Britain, Connecticut
  - Site 14, Waterbury, Connecticut
  - Site 25, Aventura, Florida
  - Site 26, Aventura, Florida
  - Site 51, Clearwater, Florida
  - Site 71, Clearwater, Florida
  - Site 61, Daytona Beach, Florida
  - Site 75, Gainesville, Florida
  - Site 33, Pensacola, Florida
  - Site 21, Stuart, Florida
  - Site 82, Tampa, Florida
  - Site 9, Venice, Florida
  - Site 83, West Palm Beach, Florida
  - Site 40, Alpharetta, Georgia
  - Site 90, Alpharetta, Georgia
  - Site 23, Atlanta, Georgia
  - Site 8, Atlanta, Georgia
  - Site 60, Powder Springs, Georgia
  - Site 55, Savannah, Georgia
  - Site 76, Boise, Idaho
  - Site 64, Champaign, Illinois
  - Site 58, Chicago, Illinois
  - Site 72, Chicago, Illinois
  - Site 74, Chicago, Illinois
  - Site 50, Evansville, Indiana
  - Site 52, Baton Rouge, Louisiana
  - Site 65, Mandeville, Louisiana
  - Site 73, Metarie, Louisiana
  - Site 15, Lutherville, Maryland
  - Site 43, Ann Arbor, Michigan
  - Site 12, Chaska, Minnesota
  - Site 80, Chesterfield, Missouri
  - Site 16, Kansas City, Missouri
  - Site 19, Kansas City, Missouri
  - Site 3, St Louis, Missouri
  - Site 17, Billings, Montana
  - Site 36, Lincoln, Nebraska
  - Site 7, Las Vegas, Nevada
  - Site 28, Reno, Nevada
  - Site 39, New Bern, North Carolina
  - Site 79, Raleigh, North Carolina
  - Site 46, Winston-Salem, North Carolina
  - Site 59, Winston-Salem, North Carolina
  - Site 45, Cincinnati, Ohio
  - Site 81, Cincinnati, Ohio
  - Site 53, Columbus, Ohio
  - Site 34, Mayfield Heights, Ohio
  - Site 78, Mogadore, Ohio
  - Site 77, Tulsa, Oklahoma
  - Site 13, Portland, Oregon
  - Site 89, Portland, Oregon
  - Site 84, Philadelphia, Pennsylvania
  - Site 63, Pottstown, Pennsylvania
  - Site 22, Warwick, Rhode Island
  - Site 24, Greenville, South Carolina
  - Site 67, Hilton Head, South Carolina
  - Site 10, Chattanooga, Tennessee
  - Site 88, Memphis, Tennessee
  - Site 56, Nashville, Tennessee
  - Site 86, Bryan, Texas
  - Site 20, Corpus Christi, Texas
  - Site 11, Houston, Texas
  - Site 30, San Antonio, Texas
  - Site 41, San Antonio, Texas
  - Site 49, Salt Lake City, Utah
  - Site 47, Charlottesville, Virginia
  - Site 2, Norfolk, Virginia
  - Site 29, Richmond, Virginia
  - Site 48, Richmond, Virginia
  - Site 42, Virginia Beach, Virginia
  - Site 5, Seattle, Washington
  - Site 38, Spokane, Washington
  - Site 32, Tacoma, Washington
- Canada (25):
  - Site 120, Abbotsford, British Columbia
  - Site 100, North Vancouver, British Columbia
  - Site 135, Victoria, British Columbia
  - Site 116, West Vancouver, British Columbia
  - Site 122, Winnipeg, Manitoba
  - Site 93, Winnipeg, Manitoba
  - Site 111, St. John's, Newfoundland and Labrador
  - Site 109, Burlington, Ontario
  - Site 114, Corunna, Ontario
  - Site 95, Hamilton, Ontario
  - Site 115, Kingston, Ontario
  - Site 107, London, Ontario
  - Site 106, Newmarket, Ontario
  - Site 137, Ottawa, Ontario
  - Site 117, Peterborough, Ontario
  - Site 113, Sarnia, Ontario
  - Site 92, Sarnia, Ontario
  - Site 96, Strathroy, Ontario
  - Site 112, Montreal, Quebec
  - Site 103, Rimouski, Quebec
  - Site 119, Sainte-Foy, Quebec
  - Site 94, Sainte-Foy, Quebec
  - Site 91, Shawinigan, Quebec
  - Site 105, Sherbrooke, Quebec
  - Site 136, Sherbrooke, Quebec
- Russia (12):
  - Site 124, Moscow
  - Site 125, Moscow
  - Site 126, Moscow
  - Site 128, Moscow
  - Site 129, Moscow
  - Site 130, Moscow
  - Site 132, Moscow
  - Site 133, Moscow
  - Site 127, Saint Petersburg
  - Site 131, Saint Petersburg
  - Site 134, Saint Petersburg
  - Site 138, Saint Petersburg